CLINICAL TRIAL: NCT01968694
Title: Effects of Intravenous Lidocaine on Endometriosis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Antje Barreveld, MD, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P002903
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Endometriosis
Keywords: endometriosis; chronic pain; intravenous lidocaine
MeSH Terms: conditions — Endometriosis; Chronic Pain | interventions — Lidocaine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Lidocaine (Experimental): IV lidocaine dosed at 8mg/kg IV (maximum 500 mg) and infused over 30 minutes
  Interventions: Drug: IV Lidocaine
- IV diphenhydramine (Placebo Comparator): IV diphenhydramine 50mg total dosed as a 10mg IV bolus and then 40mg IV infusion over 30 minutes
  Interventions: Drug: IV diphenhydramine

INTERVENTIONS:
Drug: IV Lidocaine
  Arms: IV Lidocaine
Drug: IV diphenhydramine
  Arms: IV diphenhydramine

SUMMARY:
We are doing this research study to find out if intravenous (in your vein, "IV") lidocaine can lessen pain from endometriosis. The U.S. Food and Drug Administration (FDA) has approved intravenous lidocaine to treat irregular heart beats, but the FDA has not approved intravenous lidocaine to treat pain from endometriosis. Intravenous lidocaine has been used for more than 25 years to treat different acute and chronic pain conditions but has not yet been studied for endometriosis pain.

This is a cross-over trial over two months where one month you will receive the active medication (lidocaine) and one month you will receive the active placebo (diphenhydramine, commonly known as benadryl). We will compare the effect on pain from endometriosis of lidocaine to active placebo.

ELIGIBILITY:
Inclusion criteria:

* Reproductive age women ages 18 - 50
* Endometriosis diagnosed laparoscopically or by primary care physician or gynecologist using clinical criteria
* Pain for > 6 months
* Pain most intense around time of menstrual cycle. Pain at least 5 on a 0-10 scale.
* Receiving regular monthly menses (cannot be receiving Depo-provera injections)

Exclusion criteria:

* Pregnant or breastfeeding
* On lupron therapy
* History of myocardial infarction or cardiac arrhythmias including Wolff-Parkinson-White, severe sinoatrial, atrioventricular or intraventricular heart block in the absence of a pacemaker
* History of seizure disorder
* Significant anxiety, psychosis or other cognitive disorder limiting completion of study procedures
* History of alcohol or substance abuse
* Chronic pain symptoms other than chronic pelvic pain (excluding migraine pain)
* Known hypersensitivity to amide type anesthetics
* Known hypersensitivity to diphenhydramine (benadryl)
* History of treatment with lidocaine or mexiletene
* Having or showing signs and symptoms of liver disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antje Barreveld, MD, Principal Investigator — Brigham and Women's Hospital, Newton-Wellesley Hospital
Locations (1):
- Brigham and Women's Hospital Pain Management Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 19 of the 20 enrolled started the study because one participant did not participate past consent.
Groups:
- IV Lidocaine Then IV Diphenhydramine: IV lidocaine dosed at 8mg/kg IV (maximum 500 mg) and infused over 30 minutes.
  IV diphenhydramine 50mg total dosed as a 10mg IV bolus and then 40mg IV infusion over 30 minutes.
- IV Diphenhydramine Then IV Lidocaine: IV diphenhydramine 50mg total dosed as a 10mg IV bolus and then 40mg IV infusion over 30 minutes.
  IV lidocaine dosed at 8mg/kg IV (maximum 500 mg) and infused over 30 minutes.
Period: Visit 1 (1 Day)
Arm/Group | IV Lidocaine Then IV Diphenhydramine | IV Diphenhydramine Then IV Lidocaine
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Washout (1 Month)
Arm/Group | IV Lidocaine Then IV Diphenhydramine | IV Diphenhydramine Then IV Lidocaine
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Visit 2 (1 Day)
Arm/Group | IV Lidocaine Then IV Diphenhydramine | IV Diphenhydramine Then IV Lidocaine
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Lidocaine Then IV Diphenhydramine | IV Diphenhydramine Then IV Lidocaine | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Scale (VAS)
Description: Visual Analogue Scale (VAS) ranges from 0 (no pain) to 10 (the worse imaginable pain).
  Change scores are calculated from baseline (pre-infusion) at 15 minutes after start of infusion, 30 minutes after start of infusion, and 30 minutes after infusion complete:
  (15 minutes after start of infusion value - BL pre-infusion value) (30 minutes after start of infusion value - BL pre-infusion value) (30 minutes after infusion complete value - BL pre-infusion value)
Time Frame: 15 minutes after start of infusion, 30 minutes after start of infusion, and 30 minutes after infusion complete from BL (pre-infusion)
Population: 2 participants in the IV Lidocaine arm are missing VAS 30 minutes after infusion started.
  3 participants in the IV Lidocaine arm are missing VAS 30 minutes after infusion complete.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Lidocaine | IV Diphenhydramine
Number analyzed (Participants) | 18 | 19
units on a scale
  15 minutes after start of infusion change | -2.6 [-4.5 to -0.8] | -0.2 [-1.0 to 0]
  30 minutes after start of infusion change: number analyzed (Participants) | 17 | 19
  30 minutes after start of infusion change | -3.5 [-5.0 to -2.3] | -1.5 [-2.7 to -0.1]
  30 minutes after infusion complete change: number analyzed (Participants) | 15 | 19
  30 minutes after infusion complete change | -3.6 [-4.6 to -0.6] | -1.7 [-2.7 to 0]

2. Secondary Outcome: Change in Short Form McGill Pain Questionnaire 2
Description: Short-form McGill Pain Questionnaire version 2 consists of 22 pain items (Throbbing, Shooting, Stabbing, Sharp, Cramping, Gnawing, Hot-burning, Aching, Heavy, Tender, Splitting, Tiring-exhausting, Sickening, Fearful, Punishing-cruel, Electric-shock, Cold-freezing, Piercing, Pain caused by light touch, Itching, Tingling or 'pins and needles', and Numbness). Each item is rated on a scale from 0-10, where 0=none, and 10=worst possible pain. The total pain score is the sum of these 22 items, ranging from 0-220.
  Change scores are calculated from baseline (pre-infusion) at 30 minutes, 1 week, and 1 month post-treatment:
  (30 minutes post-treatment value - BL pre-infusion value)
  (1 week post-treatment value - BL pre-infusion value)
  (1 month post-treatment value - BL pre-infusion value)
Time Frame: 30 minutes, 1 week, and 1 month post-treatment from BL (pre-infusion)
Population: 1. participant in the IV diphenhydramine arm is missing SFMPQ total score 1 week post-treatment.
  2. participants in the IV diphenhydramine arm are missing SFMPQ total score 1 month post-treatment.
  3. participants in the IV Lidocaine arm are missing SFMPQ total score 1 month post-treatment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Lidocaine | IV Diphenhydramine
Number analyzed (Participants) | 18 | 19
units on a scale
  30 minutes change from BL | -14.5 [-46 to -8] | -15 [-30 to -4]
  1 week change from BL: number analyzed (Participants) | 18 | 18
  1 week change from BL | -18 [-43 to -4] | -17 [-30 to -6]
  1 month change from BL: number analyzed (Participants) | 15 | 17
  1 month change from BL | 4 [-35 to 24] | -18 [-26 to -11]

3. Secondary Outcome: Change in Brief Pain Inventory (BPI): Pain on Average
Description: The Pain on Average score in the Brief Pain Inventory is rated from 0-10, where 0 is no pain, and 10 is pain as bad as you can imagine.
  Change scores are calculated from baseline (pre-infusion) at 1 day, 1 week, and 1 month post-treatment:
  (1 day post-treatment value - BL pre-infusion value)
  (1 week post-treatment value - BL pre-infusion value)
  (1 month post-treatment value - BL pre-infusion value)
Time Frame: 1 day, 1 week, and 1 month post-treatment from BL (pre-infusion)
Population: In the IV diphenhydramine arm 1 pt is missing BPI avg pain score at 1 week, and 2 are missing scores at 1 month. In the IV Lidocaine arm 1 pt is missing a score at 1 day, 1 is missing a score at 1 week, and 4 are missing scores at 1 month.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Lidocaine | IV Diphenhydramine
Number analyzed (Participants) | 17 | 19
units on a scale
  1 day change from BL | -2 [-3 to 0] | 0 [-2 to 1]
  1 week change from BL: number analyzed (Participants) | 17 | 18
  1 week change from BL | -2 [-2 to 0] | 0 [-1 to 0]
  1 month change from BL: number analyzed (Participants) | 14 | 17
  1 month change from BL | -1 [-2 to 0] | -1 [-1 to 1]

4. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS)
Description: The Hospital Anxiety and Depression Scale (HADS) consists of 14 items rated from 0-3 and 2 subscales Depression (7 items) and Anxiety (7 items). A higher score on each item represents more of each symptom (i.e., more depression or more anxiety). Each subscale score is the sum of the 7 items from each subscale.
  A score of 0-7 = Normal, 8-10=Borderline abnormal (borderline case), and 11-21=Abnormal (case).
  Change scores are calculated from baseline (pre-infusion) at 1 day, 1 week, and 1 month post-treatment:
  (1 day post-treatment value - BL pre-infusion value)
  (1 week post-treatment value - BL pre-infusion value)
  (1 month post-treatment value - BL pre-infusion value)
Time Frame: 1 day, 1 week, and 1 month post-treatment from BL (pre-infusion)
Population: In the IV diphenhydramine arm 1 pt is missing HADS scores at 1 week, and 3 pts are missing scores at 1 month. In the IV Lidocaine arm 3 pts are missing HADS scores at 1 month.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Lidocaine | IV Diphenhydramine
Number analyzed (Participants) | 18 | 19
units on a scale
  Anxiety 1 day change | -1 [-2 to 0] | 0 [-2 to 0]
  Anxiety 1 week change: number analyzed (Participants) | 18 | 18
  Anxiety 1 week change | -1 [-2 to -1] | -2 [-3 to 0]
  Anxiety 1 month change: number analyzed (Participants) | 15 | 16
  Anxiety 1 month change | 0 [-2 to 0] | -1.0 [-2.5 to 0]
  Depression 1 day change | -0.5 [-2.0 to 0] | 0 [-2 to 0]
  Depression 1 week change: number analyzed (Participants) | 18 | 18
  Depression 1 week change | -1 [-2 to -1] | -2 [-3 to 0]
  Depression 1 month change: number analyzed (Participants) | 15 | 16
  Depression 1 month change | -1 [-2 to 0] | -0.5 [-3 to 0]

ADVERSE EVENTS:
Groups:
- Washout Period After IV Lidocaine: Washout period after IV Lidocaine before IV diphenhydramine
- Washout Period After IV Diphenhydramine: Washout period after IV diphenhydramine before IV Lidocaine
Arm/Group | IV Lidocaine | IV Diphenhydramine | Washout Period After IV Lidocaine | Washout Period After IV Diphenhydramine
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes